CLINICAL TRIAL: NCT06598501
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) and Cognitive Behavioral Therapy (CBT) in the Management of Gambling Disorder in Indonesia: a Pilot and Feasibility Study
Brief Title: Repetitive Transcranial Magnetic Stimulation (rTMS) and Cognitive Behavioral Therapy (CBT) for Gambling Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Kristiana Siste, Dr. dr. Kristiana Siste, SpKJ(K) - Head of Department of Psychiatry, Faculty of Medicine, Indonesia University, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 34/IV/KS/05/2023
Record Dates: First submitted 2024-09-14; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Gambling Disorder
MeSH Terms: conditions — Gambling | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rTMS and CBT (Experimental): During 5 weeks of therapy, the subjects will undergo 12 CBT sessions (30-40 minutes) combined with 15 rTMS procedures (20 minutes).
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — an open arm study of 10 gambling disorder subjects will be conducted to determine the efficacy and feasibility of a multimodalistic therapy of rTMS and Cognitive Behavioral Therapy (CBT) for gambling disorder in Indonesia.

SUMMARY:
Treatment options for gambling disorder (GD) remain limited, with no pharmacotherapy proven effective. As of date, cognitive behavioral therapy (CBT) is the preferred therapy for GD, but the improvements often require months to show, highlighting the need for a more comprehensive therapy. Repetitive transcranial magnetic stimulation (rTMS) is a promising treatment modality in alleviating craving. Studies have shown potential benefit of combining both CBT and rTMS in substance addiction, but not in GD. Thus, this study aims to determine the feasibility and efficacy of rTMS and CBT combination therapy in the management of GD in Indonesia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with pathological gambling (SOGS score ≥ 5)
* Subjects aged 18-70 years old
* Subjects who understand Bahasa Indonesia
* Subjects who agree to participate and receive treatment

Exclusion Criteria:

* Subjects with history of psychotic disorder and personality disorder according to ICD-11
* Subjects with severe neurological disorder comorbidities, which cause seizure or loss of consciousness
* Subjects with intellectual disability
* Subjects with history of neurostimulation
* Subjects with history of medical implant
* Subjects currently or expecting pregnancy
* Subjects fulfilling diagnostic criteria of substance use disorder in the last 6 months

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Improvement in pathological gambling score | Baseline (week 0), interim assessment (week 3), post-intervention (week 6), follow up at 3 months and 6 months after intervention
  South Oaks Gambling Screen (SOGS), Indonesian version, with minimum score of 0 and maximum score of 20. A score of 0-2 indicates no pathological gambling; a score of 3-4 indicates problems with gambling, and a score of 5 or more indicates that the subject is a probable pathological gambler. Lower score indicates a better outcome.
Improvement in gambling symptoms severity | Baseline (week 0), interim assessment (week 3), post-intervention (week 6), follow up at 3 months and 6 months after intervention
  Gambling Symptoms Assessment Scale (G-SAS), Indonesian version, with minimum score of 0 and maximum score of 48. Interpretations: Mild (8-20), Moderate (21-30), Severe (31-40), and Extreme (41-48). Lower score indicates a better outcome.
Improvement in gambling urge | Baseline (week 0), interim assessment (week 3), post-intervention (week 6), follow up at 3 months and 6 months after intervention
  Gambling Urge Scale (GUS), Indonesian version, with minimum score of 0 and maximum score of 42. Lower score indicates a better outcome.
Improvement in gambling related cognitive distortions | Baseline (week 0), interim assessment (week 3), post-intervention (week 6), follow up at 3 months and 6 months after intervention
  Gambling Related Cognitions Scale (GRCS), Indonesian version, with 5 cognitive distortion domains. Lower score indicates a better outcome.

SECONDARY OUTCOMES:
Improvement in gambling-related cognitive functions | Baseline (week 0), interim assessment (week 3), post-intervention (week 6), follow up at 3 months and 6 months after intervention
  Creyos (formerly Cambridge Brain Sciences, CBS), measures 12 domains of cognitive function with the subject results compared with their respective average age results in percentile. A higher percentile is a better outcome.
Improvement in depression symptoms | Baseline (week 0), post-intervention (week 6), follow up at 3 months and 6 months after intervention
  Beck Depression Inventory-II (BDI II), measures severity of depression symptoms, with minimum score of 0 and maximum score of 63. Interpretation: (1) minimal (0-13), (2) mild (14-19), (3) moderate (20-28), and (4) severe (29-63). Lower score indicates a better outcome.
Improvement in self-reported psychological distress | Baseline (week 0), post-intervention (week 6), follow up at 3 months and 6 months after intervention
  20-item Self-Reporting Questionnaire (SRQ-20), Indonesian version, measures non-specific psychological distress. Score range 0-20, with scores >10 classified as mental distress. Lower score indicates a better outcome.
Improvement of overall severity of illness | Baseline (week 0), interim assessment (week 3), post-intervention (week 6), follow up at 3 months and 6 months after intervention
  Clinical Global Impression (CGI), measure overall severity of illness and improvement observed by the clinician. Lower score indicates a better outcome.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Siste K, Sen LT, Murtani BJ, Hanafi E, Kusuma KS, Aryani A, Schellekens A, van Eijndhoven P, Dalhuisen I, Biemans T. Utilizing repetitive transcranial magnetic stimulation in the management of gambling disorder in Indonesia: protocol for a pilot and feasibility study. Front Psychiatry. 2025 Sep 5;16:1658195. doi: 10.3389/fpsyt.2025.1658195. eCollection 2025. PMID 40980053